CLINICAL TRIAL: NCT06253507
Title: A Phase I/II, Non-Randomized, Open-Label Study of pCCLCHIM-p47 (Lentiviral Vector Transduced CD34+ Cells) in Patients With p47 Autosomal Recessive Chronic Granulomatous Disease (AR-CGD)
Brief Title: pCCLCHIM-p47 (Lentiviral Vector Transduced CD34 Plus Cells) in Patients With p47 Autosomal Recessive Chronic Granulomatous Disease (AR-CGD)
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001562; 001562-I
Record Dates: First submitted 2024-02-09; First posted 2024-02-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01-08

CONDITIONS: p47; Autosomal Recessive; Chronic Granulomatous Disease
Keywords: p47 Phox; Autosomal Recessive; Chronic Granulomatous Disease; Gene Therapy; Lenti Vector
MeSH Terms: conditions — Granulomatous Disease, Chronic; Granulomatous Disease, Chronic, Autosomal Recessive, Cytochrome B-Positive, Type I

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Biological: Cryopreserved Autologous CD34+ cells transduced with pCCLCHIM-p47

INTERVENTIONS:
Biological: Cryopreserved Autologous CD34+ cells transduced with pCCLCHIM-p47 — Cryopreserved autologous CD34+ cells transduced ex vivo with the pCCLCHIM-p47 vector containing the human p47phox (NCF1) gene in final formulation and container closure system, ready for intended medical use.
  The minimum cell dose for infusion is 3 x 10^6 CD34+/kg.

SUMMARY:
Background:

Chronic granulomatous disease (CGD) is a genetic disorder. People with CGD are missing a gene that affects their white blood cells. White cells are part of the immune system, and people with GCD are vulnerable to many infections. Researchers want to test a new treatment to replace the missing gene that may be safer than the current treatment for CGD.

Objective:

To test a new type of gene therapy in people with CGD.

Eligibility:

People aged 3 years or older with CGD.

Design:

Participants will undergo apheresis: Blood will be collected through a tube attached to a needle inserted in a vein; the blood will run through a machine that separates certain cells (stem cells); the remaining blood will be returned to the body through a second needle. The participant s stem cells will be modified in a laboratory to add the gene they are missing.

Participants will stay in the hospital for about 40 days.

For the first 10 days, they will undergo many exams, including imaging scans and tests of their heart and lung function. They will receive drugs to prepare their bodies for the gene therapy. They will receive a "central line": A hollow tube will be inserted into a vein in the chest, with a port opening above the skin. This port will be used to draw blood and administer drugs without the need for new needle sticks.

For the gene therapy, each participant s own modified stem cells will be put into their body through the port.

Participants will have 8 follow-up visits over 3 years.

DETAILED DESCRIPTION:
Study Description:

This is a phase I/II, non-randomized, open-label study of a single infusion of autologous CD34+ cells transduced ex vivo with pCCLCHIM-p47 in 5 patients with p47-AR CGD conditioned with high dose busulfan.

Objectives:

Primary Objectives:

To evaluate the efficacy of pCCLCHIM-p47 transduced autologous CD34+ cells treatment in p47 AR-CGD patients as measured by engraftment of genetically modified cells at 6 months.

Secondary Objectives:

* Safety
* Long term engraftment (assessments at 1 year, 2 years, and 3 years)
* Event Free Survival
* Clinical Efficacy and Health Assessment

Exploratory Objectives:

* Assessment of biomarker utility
* Evaluation of the human microbiome during pCCLCHIM-p47 gene therapy.
* Patient reported assessment of efficacy (QOL)

Endpoints:

Primary Endpoint of this study will be engraftment of genetically modified cells as defined by presence of >10% oxidase positive cells at 6 months.

* Secondary Endpoints will consist of:
* Safety: assessed by recording of the incidence of adverse events.

  * Record clinical adverse events and clinically significant laboratory abnormalities.
  * Evaluate overall incidence of adverse events for the study as a whole.
  * Monitor the incidence of serious adverse events.
  * Measure overall survival at 3 years post-transplant
  * Assessment of vector safety by vector insertion site analysis (VISA) and replication competent lentivector (RCL) testing.
* Long term multilineage engraftment, as measured by:

  * Expression of p47 phox in neutrophils at 6, 12, 18, 24, and 36 months.
  * Hematological reconstitution by 90 days post treatment (absolute neutrophil count >500 cells/microliter on three consecutive samples over at least ten days).
  * NADPH Oxidase activity in monocytes by dihydrorhodamine (DHR) flow cytometry at 6, 12, 18, 24, and 36 months.
  * Percentage of gene modified CD34+ hemopoietic cells in BM at 6, 12, 18, 24, 30, and 36 months as assessed by vector copy number (VCN) qPCR.
  * VCN in cell lineages present in PB cells at months 1, 3, 6, 9, 12, 18, 24, and 36.
* Event free Survival

  * Resolution of either underlying inflammation and/or infection related to P47 deficiency without recurrence for 3 years.
  * Rate of severe (as defined by CTCAE v 5.0 - grade 3 to 5) CGD related infections after withdrawal of antimicrobial prophylaxis in time periods 6-12 and 6-36 months post treatment.
* Assessment of clinical efficacy and health by:

  * The nutritional status (height, weight, serum albumin) at 36 months.
  * Growth and development of pediatric subjects at 36 months.
  * Frequency of severe infections (days requiring IV antibiotics and/or hospitalization for treatment) at 36 months.
  * Presence of inflammatory complications (days requiring hospitalizations) at 36 months.

Tertiary Endpoints:

* Utility of Biomarker assessment
* Stool collection for microbiome analysis (optional)
* Patient Quality of life questionnaire collection

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

-Must have confirmed genetic diagnosis of p47 AR-CGD by identification of a mutation in the responsible genes or protein analysis demonstrating lack of P47 expression and supported by laboratory evidence for absent or reduction > 95% of the biochemical

activity of the NADPH-oxidase.

* Must weigh at least 15 kg.
* Adult Patient must be willing to sign and date informed consent form.
* Parent/guardian must be willing to sign and date informed consent form for child and where appropriate, child may sign assent.
* State willingness to comply with all study procedures and availability for the duration of the study.
* Male or female must be at least 3 years of age.
* Do not have an appropriately HLA matched donor (related or unrelated)
* Must have had at least a history of a prior CGD related infection and/or an ongoing/refractory severe infection requiring hospitalization and/or inflammatory complications requiring hospitalization despite conventional therapy.
* Patients will be collected as per standard of care mobilization and apheresis procedures as performed at the Clinical Center. Patients will have consented onto the gene therapy study prior to collection; however products collected prior to the study for other protocols may be used as part of the back up.

  * Patient must weigh at least 15 kilograms body weight.
  * Normal female donors of childbearing potential may be entered if using effective contraception and having a negative serum pregnancy test within one week of beginning G-CSF administration.
* Ability to take oral medication and be willing to adhere to the prophylactic regimen.
* For females of reproductive potential, must agree to use 2 forms of highly effective contraception throughout study participation (for a minimum of 3 months after having received the genetically modified cells but preferably for the first 2 years.)

  * For females (will be counseled on appropriate combinations for best efficacy):

    * Condoms, male or female, with or without a spermicide.
    * Diaphragm or cervical cap with spermicide.
    * Intrauterine device.
    * Contraceptive pills or patch, Norplant, Depo-Provera, or other FDAapproved contraceptive method.
    * Having a male partner who has previously undergone a vasectomy.
  * For males of reproductive potential: use of condoms or other methods to ensure effective contraception prevention with partner.
* Agreement to adhere to Lifestyle Considerations throughout study duration.
* Must provide a durable power of attorney (DPA) for health care decisions to an appropriate adult relative or guardian in accordance to NIH-200 "NIH Advance Directive for Health Care and Medical Research Participation".
* All patients must be willing to allow storage of blood samples for gene therapy studies.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Patient/Parent/Guardian unable or unwilling to comply with the protocol requirements.
* Contraindication for leukapheresis (anemia Hb <8g/dL, cardiovascular instability, severe coagulopathy, uncontrolled seizure disorder).
* Pregnancy or lactation.
* Tested positive (definitive) for the presence of multiple types (2 or more) of anti-platelet antibodies.
* Patient will be excluded if they have any of the following within 8 weeks of entering the trial.

  * Hematologic

    * Anemia (hemoglobin < 8 g/dL).
    * Neutropenia (absolute granulocyte count <1,000/mm3)
    * Thrombocytopenia (platelet count < 100,000/mm3).
    * Prothrombin Time (PT) or Partial thromboplastin time (PTT) > 2 X the upper limits of normal (ULN) (Patients with a correctable deficiency controlled on medication will not be excluded).
    * Cytogenetic abnormalities known to be associated with hematopoietic defect on peripheral blood or bone marrow.
  * Infectious

    ---Evidence of infection with HIV-1 and -2, or active Hepatitis B, Hepatitis C, Adenovirus, Parvovirus, Toxoplasmosis, or any other uncontrolled viral infection.
  * Pulmonary

    ---Resting O2 saturation by pulse oximetry < 90% on room air.
  * Cardiac

    * Ejection fraction by Echocardiogram of less than 40%

OR

---Uncorrected congenital cardiac malformation with clinical symptomatology

OR

* Abnormal EKG which with additional work up (including a Cardiology consult) indicates cardiac pathology incompatible with the use of high dose busulfan.

  --Hepatic
* Transaminases >5X upper limit of normal.

  * General

    * Expected survival < 6 months.
    * Major congenital anomaly.
    * Contraindication for administration of conditioning medication.
    * Current or active malignancy or prior hematologic malignancy.
    * Uncontrolled hypertension (systolic greater than 1 SD of the mean expected for age despite adequate medication).
    * Uncontrolled tachycardia with resting heart rate greater than 1 standard deviation for age group despite medications.
    * Neurologic deficits determined to interfere with ability to comply with study interventions.
  * Known serious or anaphylactic allergic reactions to components of the Busulfan or to DMSO.
  * Treatment with another investigational drug or other intervention within 6 months.
  * Unable to undergo apheresis:

    * Patients who are hemodynamically unstable (systolic or diastolic blood pressure fall of 20 mm Hg from the stable patient s baseline measurement) or requiring mechanical respiratory assistance are excluded.
    * History of vasculitis or any illness that precludes apheresis as defined by the Cellular Engineering Department.
  * Administration of gamma-interferon within 30 days before the infusion of transduced, autologous CD34+ cells.
  * Acute infection diagnosed but not treated at time of enrollment. Patients will be delayed for enrollment until infection has resolved or if not resolving with adequate standard medical care, the patient will then be re-eligible for treatment as this would have them meeting the inclusion criteria of a refractory infection. (Patients that develop an infection during the conditioning [after enrollment and having started the busulfan] will proceed with the study.)
  * Any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the patient or would preclude the patient from successful study completion.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of pCCLCHIM-p47 transduced autologous CD34+ cells treatment in p47 AR-CGD patients as measured by engraftment of genetically modified cells. | 6 months to 1 year.

SECONDARY OUTCOMES:
Safety | Length of study
  assessed by recording of the incidence of adverse events for the study as a whole
Long term Engraftment | 6, 12, 18, 24, and 36 months
Event Free Survival | 3 years
Clinical Efficacy and Health Assessment | 24 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Kang, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001562-I.html